CLINICAL TRIAL: NCT07008729
Title: Heart Failure Patient Management and Interventions Using Continuous Patient Monitoring Outside Hospitals and Real-world Data
Acronym: RETENTION
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Puerta de Hierro University Hospital (Other)
Collaborators: Hannover Medical School (Other); Attikon Hospital (Other); IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other); Onassis Cardiac Surgery Centre (Other); Hospital Universitario Ramon y Cajal (Other)
Responsible Party: Principal Investigator, Mercedes Rivas-Lasarte, Principal Investigator, MD PHD, Cardiology Department, Puerta de Hierro University Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: H2020-SC1-BHC-2018-2020 GA 965; PI 152/22 (Other: HOSPITAL PUERTA DE HIERRO)
Record Dates: First submitted 2025-05-13; First posted 2025-06-06 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Chronic Heart Failure; Heart Transplant Recipient; Left Ventricular Assist Device
Keywords: Remote patient management; Telemonitoring; Chronic heart failure; Heart transplant; durable left ventricular assist device; hospitalisations; heart failure decompensation

STUDY DESIGN:
Who Masked: Participant, Care Provider
Masking Description: The care providers will be masked to the data collected by the control group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): The RETENTION platform will offer to the clinician in the experimental arm all the data gathered by the devices (smart watch, scale, oximeter, blood pressure monitor, temperature, medication adherence, weather and pollution indexes). along with artificial intelligence recommendations.
  Interventions: Device: Heart monitoring tools (data revision)
- Control group (Placebo Comparator): Patients in the control group will be monitored but the data will not be available to the clinicians nor the artificial intelligence recommendations.
  Interventions: Other: Control (Standard treatment)

INTERVENTIONS:
Device: Heart monitoring tools (data revision) — data collected by the devices will be reviewed by the treating physician in the intervention group
  Arms: Intervention group
Other: Control (Standard treatment) — Patients in the control group will be monitored but the information will not be available for the clinicians nor the artificial intelligence recommendations
  Arms: Control group

SUMMARY:
The goal of this study is to create a digital platform for managing patients with chronic heart failure, those with long-term ventricular assistance, or heart transplant recipients. This platform aims to help doctors make clinical decisions and change treatments based on continuous monitoring and the collection of medical, clinical, physiological, behavioral, psychosocial, and real-world data from these patients.

The ultimate goal is to reduce mortality and hospitalization rates for this group of patients while improving their quality of life, safety, and well-being.

To do this, participants will be divided into two groups:

* Intervention Group: The data collected by the platform will be available to their treating doctors.
* Control Group: Doctors will not have access to the data.

All participating patients will receive a set of devices and sensors to collect data such as vital signs, physical activity, sleep quality, psychological and nutritional status, and environmental data. All this information will be gathered through a mobile app designed for the study.

The follow-up will last for 18 months, during which there will be 4 in-person medical visits (spaced 4 months apart). Participation in the study won't affect patients' scheduled medical visits related to their illness or their usual treatment.

DETAILED DESCRIPTION:
Specifically, the devices that will be given to the patients and their required use will be as follows:

A Smartphone: This will have the app with the platform designed for the study. The patient must interact with it daily to enter data.

A Blood Pressure Monitor: The patient will need to take their blood pressure every day and send it via Bluetooth to the mobile platform (the connection setup will be done by the study team before giving it to the patients).

An Oxygen Saturation Monitor: The patient will need to check their oxygen levels daily and send the data via Bluetooth to the mobile platform (the connection setup will be done by the study team before giving it to the patients).

A Scale: The patient will need to weigh themselves daily and transmit the data via Bluetooth to the mobile platform (the connection setup will be done by the study team before giving it to the patients).

A Smartwatch: The patient must send data on their physical activity and sleep daily via Bluetooth to the mobile platform (the connection setup will be done by the study team before giving it to the patients).

Home Humidity and Temperature Sensors and a Home Gateway Device (Raspberry Pi): The patient will need to connect this last device to their home internet network. The connection setup will be done by the study team before giving it to the patients.

There are other data and information that the patient must manually enter into the app, such as daily body temperature, symptoms they experience (like increased fatigue or shortness of breath), or data on the functioning of the long-term ventricular assistance (controller parameters or alarm presence). Additionally, the app will show the patient's current medication, which they need to confirm they have taken correctly.

The scheduled visits during the study will take place at the Baseline and every four months. These visits will include an in-person medical visit, an electrocardiogram, a blood test, and a 6-minute walk test. Also, at each visit, a series of questionnaires will be given to assess the patient's cognitive, nutritional, and psychological state, as well as their quality of life and that of their primary caregivers. Some visits will also include more specific cardiac tests, like an echocardiogram or a cardiopulmonary exercise test.

If during the study follow-up, the treating doctors unexpectedly discover any information that affects the patient's health or quality of life, the patient will be informed immediately, even if it is unrelated to the study's purpose.

All data recorded throughout the study will be stored anonymously by the study platform.

ELIGIBILITY:
Inclusion Criteria:

* Age of 18-75 years.
* Ability to understand and provide consent in order to participate in the study.
* Have a cognitive assessment score of > 22 as assessed by the Montreal Cognitive Assessment (MoCA), ( adults without or with mild cognitive impairment at most).
* Have a depression score as assessed by Personal Health Questionnaire-9 (PHQ-9) score < 10.
* Provide written informed consent.
* For Heart Failure patients: 1) have a diagnosis of symptomatic heart failure (class II or III according to the New York Heart Association Classification); 2) have echocardiographically determined left ventricular ejection fraction (LVEF) ≤40%; 3) have been hospitalized due to cardiovascular reasons or had urgent visit to the Emergency Department due to decompensated HF that required administration of intravenous diuretics within the last 12 months before randomization (Currently hospitalized patients can be included provided they do not fulfill exclusion criterion of being currently with in-hospital administration of IV diuretics/vasoactive/inotropic drugs).
* For patients with ventricular assist devices (VAD): have left ventricular assist device (LVAD) implanted either as destination therapy or as bridge-to-transplantation, within at least 90 days and no longer than 48 months before randomization
* for heart transplant recipients: have been discharged following heart transplantation within at least 30 days and no longer than 36 months before study randomization.

Exclusion Criteria:

* Is clinically unstable at the time of randomization as defined by: administration of intravenous diuretics during the last 12 hours or intravenous vasodilators or inotropes during the last 48 hours before randomization.
* Has acute coronary syndrome within the last 30 days before randomization.
* Has acute inflammatory heart disease, (for instance, acute myocarditis), within 90 days prior to randomization.
* Has a planned revascularisation, cardiac resynchronization therapy (CRT) implantation or any valvular procedures within 3 months after randomization
* Has known current alcohol or illicit drug abuse.
* Shows significant impairment or unwillingness to use the telemonitoring equipment (for instance, dementia, impaired self-determination, lacking ability to communicate).
* Has any severe non-cardiovascular disease limiting life expectancy to less than 1 year.
* Is pregnant.
* Participates currently in other telemonitoring programs/studies using smart devices

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 390 (Actual)
Dates: Start 2024-04-24 (Actual); Primary Completion 2026-08-31 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
Difference in days lost due to unplanned cardiovascular hospitalizations or all-cause death between groups | From the enrollment to the end of the follow up (18 months)
  Comparison of days lost due to unplanned cardiovascular hospitalizations or all-cause death between groups
Differences in the rates of occurrence of death or unplanned hospitalization/ambulatory administration of intravenous (iv) diuretics, iv antibiotics or iv steroids | From the enrollment to the end of the follow up (18 months)
  Comparison of the rates of the occurrence of death or unplanned hospitalization/ambulatory administration of intravenous (iv) diuretics, iv antibiotics or iv steroids between groups

SECONDARY OUTCOMES:
Rates of all-cause mortality | From the enrollment to the end of the follow up (18 months)
Rates of cardiovascular mortality | From the enrollment to the end of the follow up (18 months)]
Differences in time to first unplanned HF hospitalization | From the enrollment to the end of the follow up (18 months)]
Differences in time to first unplanned cardiovascular hospitalization | From the enrollment to the end of the follow up (18 months)]
Rate of total unplanned HF hospitalizations | From the enrollment to the end of the follow up (18 months)
Rate of total unplanned cardiovascular hospitalizations | From the enrollment to the end of the follow up (18 months)
Differences in days lost due to HF hospitalizations | From the enrollment to the end of the follow up (18 months)]
Differences in the number of Smart device alarm notifications | From the enrollment to the end of the follow up (18 months)
Change in Kansas City Cardiomyopathy Questionnaire (KCCQ) score | From the enrollment to the end of the follow up (18 months)
  between Baseline and last visit. KCCQ ranges from 0 to 100, higher scores indicating higher quality of life
Change in the levels of NT-proBNP | From the enrollment to the end of the follow up (18 months)
  Between Baseline and last visit
Change in the Depression Score Patient Health Questionnaire 9 (PHQ-9) | From the enrollment to the end of the follow up (18 months)
  Between baseline and last visit
Change in the Heart Failure Caregiver Questionnaire (HF-CQ version 5.0) | From the enrollment to the end of the follow up (18 months)]
  Between baseline and last visit
Difference in the rate of rejection needing treatment in heart transplant patients | From the enrollment to the end of the follow up (18 months)
Driveline infection needing antibiotic in left ventricular assist device (LVAD) patients | From the enrollment to the end of the follow up (18 months)
Differences in the rate of unplanned visit for heart failure requiring intravenous diuretics | From the enrollment to the end of the follow up (18 months)
Difference in the number of visits outside the protocol | From the enrollment to the end of the follow up (18 months)

CONTACTS AND LOCATIONS:
Overall Officials: Maria Haritou, PhD, Study Chair — ICCS
Locations (6):
- Medizinische Hochschule Hannover ('Mhh'), Hanover, Germany
- Greece (2):
  - National and Kapodistrian University of Athens, Athens
  - Onassis Cardiac Surgery Center, Athens
- Alma Mater Studiorum - Universita Di Bologna, Bologna, Italy
- Spain (2):
  - Hospital Universitario Puerta de Hierro, Majadahonda, Madrid
  - Hospital Universitario Ramón Y Cajal, Madrid

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code

REFERENCES:
- [Background] Scott IA, Scuffham P, Gupta D, Harch TM, Borchi J, Richards B. Going digital: a narrative overview of the effects, quality and utility of mobile apps in chronic disease self-management. Aust Health Rev. 2020 Feb;44(1):62-82. doi: 10.1071/AH18064. PMID 30419185
- [Background] Ski CF, Thompson DR, Brunner-La Rocca HP. Putting AI at the centre of heart failure care. ESC Heart Fail. 2020 Oct;7(5):3257-3258. doi: 10.1002/ehf2.12813. Epub 2020 Jun 17. No abstract available. PMID 32558251
- [Background] McConnell MV, Turakhia MP, Harrington RA, King AC, Ashley EA. Mobile Health Advances in Physical Activity, Fitness, and Atrial Fibrillation: Moving Hearts. J Am Coll Cardiol. 2018 Jun 12;71(23):2691-2701. doi: 10.1016/j.jacc.2018.04.030. PMID 29880130
- [Background] Dorsey ER, Yvonne Chan YF, McConnell MV, Shaw SY, Trister AD, Friend SH. The Use of Smartphones for Health Research. Acad Med. 2017 Feb;92(2):157-160. doi: 10.1097/ACM.0000000000001205. PMID 27119325
- [Background] Liu L, Stroulia E, Nikolaidis I, Miguel-Cruz A, Rios Rincon A. Smart homes and home health monitoring technologies for older adults: A systematic review. Int J Med Inform. 2016 Jul;91:44-59. doi: 10.1016/j.ijmedinf.2016.04.007. Epub 2016 Apr 19. PMID 27185508
- [Background] Goswami R. The current state of artificial intelligence in cardiac transplantation. Curr Opin Organ Transplant. 2021 Jun 1;26(3):296-301. doi: 10.1097/MOT.0000000000000875. PMID 33938466
- [Background] Shahbazi F, Asl BM. Generalized discriminant analysis for congestive heart failure risk assessment based on long-term heart rate variability. Comput Methods Programs Biomed. 2015 Nov;122(2):191-8. doi: 10.1016/j.cmpb.2015.08.007. Epub 2015 Aug 24. PMID 26344584
- [Background] Tripoliti EE, Papadopoulos TG, Karanasiou GS, Naka KK, Fotiadis DI. Heart Failure: Diagnosis, Severity Estimation and Prediction of Adverse Events Through Machine Learning Techniques. Comput Struct Biotechnol J. 2016 Nov 17;15:26-47. doi: 10.1016/j.csbj.2016.11.001. eCollection 2017. PMID 27942354
- [Background] Bennett MK, Shao M, Gorodeski EZ. Home monitoring of heart failure patients at risk for hospital readmission using a novel under-the-mattress piezoelectric sensor: A preliminary single centre experience. J Telemed Telecare. 2017 Jan;23(1):60-67. doi: 10.1177/1357633X15618810. Epub 2016 Jul 9. PMID 26670209
- [Background] Yun JE, Park JE, Park HY, Lee HY, Park DA. Comparative Effectiveness of Telemonitoring Versus Usual Care for Heart Failure: A Systematic Review and Meta-analysis. J Card Fail. 2018 Jan;24(1):19-28. doi: 10.1016/j.cardfail.2017.09.006. Epub 2017 Sep 20. PMID 28939459
- [Background] Savarese G, Lund LH. Global Public Health Burden of Heart Failure. Card Fail Rev. 2017 Apr;3(1):7-11. doi: 10.15420/cfr.2016:25:2. PMID 28785469
- [Background] Ong MK, Romano PS, Edgington S, Aronow HU, Auerbach AD, Black JT, De Marco T, Escarce JJ, Evangelista LS, Hanna B, Ganiats TG, Greenberg BH, Greenfield S, Kaplan SH, Kimchi A, Liu H, Lombardo D, Mangione CM, Sadeghi B, Sadeghi B, Sarrafzadeh M, Tong K, Fonarow GC; Better Effectiveness After Transition-Heart Failure (BEAT-HF) Research Group. Effectiveness of Remote Patient Monitoring After Discharge of Hospitalized Patients With Heart Failure: The Better Effectiveness After Transition -- Heart Failure (BEAT-HF) Randomized Clinical Trial. JAMA Intern Med. 2016 Mar;176(3):310-8. doi: 10.1001/jamainternmed.2015.7712. PMID 26857383
- See also: Oficial project's web site. It provides information about the project to every user. — https://www.retention-project.eu/